CLINICAL TRIAL: NCT03129165
Title: ProSALUTE: a New Community Program for Cardiovascular Health
Brief Title: ProSALUTE: Community Program for Cardiovascular Health
Acronym: ProSALUTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, José Pablo Werba, Head of Unit of Atherosclerosis Prevention, Principal Investigator, Specialist in Internal Medicine, Centro Cardiologico Monzino
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R212/15 - CCM 226
Record Dates: First submitted 2017-03-30; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Primary Prevention
Keywords: Cardiovascular diseases; Public Health; Hypertension; Smoking; Hypercholesterolemia; Food Habits; Exercise; Anxiety; Depression; Obesity; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Smoking; Hypercholesterolemia; Feeding Behavior; Motor Activity; Anxiety Disorders; Depression; Obesity; Diabetes Mellitus | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening and prevention of CVD (Experimental)
  Interventions: Other: Screening and prevention of CVD

INTERVENTIONS:
Other: Screening and prevention of CVD — Drug: Pharmacological control of risk factors in agreement with primary physicians.
  Behavioral: Smoking cessation / Control of depression and anxiety / Nutritional counseling / Motivation for physical activity.
  Social: Social worker care.

SUMMARY:
The purpose of this study is to determine the efficacy and cost/effectiveness (change in CV risk factors and lifestyle vs costs) of ProSALUTE as a new organizational model of primary CV prevention.

DETAILED DESCRIPTION:
Primary Cardiovascular (CV) prevention programs in the healthcare place and community-based interventions have a variable impact on health at the population level. The largest benefit may be obtained by addressing high-risk, disadvantaged and traditionally hard-to-reach groups.

Effective actions include health promotion, timely screening of modifiable risk factors, application of evidence-based targets and interventions, broad access to heart-friendly environments/facilities and dissemination of favorable social norms. Thus, community prevention is a multifaceted task that requires multidisciplinary collaboration. A suitable program should be tailored to the specific social context and make the most of local resources to improve access, adherence and continuity, as well as sustainability.

ProSALUTE is a new model of primary CV prevention for the prevalently low-income and multiethnic community of Ponte Lambro (n=3600 adults), the neighborhood where the coordinating hospital (Centro Cardiologico Monzino, Milan, Italy) is located.

Under the coordination of a Case Manager (a Nursing Researcher) the citizens are involved in a prevention program, which is personalized (content and intensity) according to the individual global risk and specific risk factors. The citizens follow an individualized schedule of short-term specialist care. Besides, the participants are "gently nudged" to make use of local resources that may contribute to sustain a healthy life-style (e.g. parks, gyms, social services, etc). Moreover, public preventive events for the community are devised (e.g. healthy-cooking course, walking groups, etc) through a collaborative network with representatives of the neighborhood.

ELIGIBILITY:
Inclusion Criteria:

* Live in Milan at neighborhood of Ponte Lambro

Exclusion Criteria:

* Patients with known atherosclerotic disease (secondary prevention)
* Severe diseases or disabilities that hinder the participation in the program

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-05-11 (Actual); Primary Completion 2018-05-11 (Estimated); Study Completion 2018-05-11 (Estimated)

PRIMARY OUTCOMES:
Primary adherence at baseline screening | Baseline
  Primary adherence evaluated as the ratio between the number of subjects enrolled and the number of subjects actively contacted through personal postal mail

SECONDARY OUTCOMES:
Influence of education level on primary adherence | Baseline
  Assessed as rate of primary adherence according to educational level (years of schooling <8, 8-12 or >12)
Influence of working category on primary adherence | Baseline
  Assessed as rate of primary adherence according to working category (manual worker, service worker, office worker, unemployed, retired)
Influence of immigrant or native status on primary adherence | Baseline
  Assessed as rate of primary adherence according to immigrant (from any country) or native status
Awareness of own cardiovascular risk factors | Baseline
  Awareness assessed as prevalence of knowledge (answer: known value or not known) of levels of the following personal cardiovascular risk factors: total cholesterol, triglycerides, glycaemia, systolic and diastolic blood pressure
Accuracy of the perception of own cardiovascular risk | Baseline
  Accuracy assessed as concordance (using Cohen's kappa test) between risk perception (evaluated through a 5 point Likert scale questionnaire: from very low to very high) and estimated cardiovascular risk (evaluated through the Framingham Risk Score)
Prevalence of positive screening for anxiety | Baseline
  Anxiety assessed using General Anxiety Disorder 2 (GAD-2) test and defined as positive with a score ≥3
Prevalence of positive screening for depression | Baseline
  Depressive mood assessed using Patient Health Questionnaire 2 (PHQ-2) test and defined as positive with a score ≥3
Extent of adherence to the Mediterranean Diet (MD) | Baseline
  Extent of adherence to MD assessed using the PREDIMED questionnaire and score, using three categories (0-7 low adherence; 8-9 medium adherence, ≥10 high adherence)
Prevalence of physically active subjects | Baseline
  Physical activity (PA) assessed using the PASSI questionnaire and physically active subjects defined according to the WHO 2010 Guidelines
Human resources utilization | Baseline
  Percent of enrolled subjects allocated to medical visit, interview with nutritionist, motivational interview to promote physical activity, smoking-cessation program, interview with psychologist
Persistence in the program at 6th months | 6 months
  Persistence assessed as the ratio between subjects followed at 6 months and subjects enrolled
Changes in adherence to MD at 6 months | 6 months
  Assessed as the net improvement in category of adherence to MD (number of those who increased minus number of those who decreased)
Changes in PA at 6 months | 6 months
  Assessed as the net improvement in category of PA level (number of sedentary subjects shifted to active or moderate minus number of active or moderate shifted to sedentary)
Changes in declared cigarette consumption | 6 months
  Assessed as the net improvement in extent of cigarette consumption (number of smokers who reduced the number of cigarettes/day minus number of smokers who increased the number of cigarettes/day)
Changes in objective measures of cigarette smoke exposure | 6 months
  Assessed as the net improvement in exhaled Carbon Monoxide (CO) (number of smokers who reduced ≥10% exhaled CO ppm minus number of smokers who increased ≥10% exhaled CO ppm)
Change in positive screening for anxiety | 6 months
  Assessed as the net improvement in screening for anxiety (number of positive who became negative minus number of negative who became positive)
Change in positive screening for depression | 6 months
  Assessed as the net improvement in screening for depression (number of positive who became negative minus number of negative who became positive)
Global change in traditional risk factors at 6th months | 6 months
  Assessed as the number of subjects who improved by ≥10% at least one traditional CV risk factor measure without worsening by ≥10% any other CV risk factor measure. The CV risk factors considered are: glycaemia >126 mg/dl, LDL-C >115 mg/dl, systolic blood pressure >140 mmHg and BMI >28
Global change in estimated risk at 6th months | 6 months
  Assessed as net improvement in Framingham Risk Score (number of subjects who reduced the score minus number of subjects who increased the score)
Persistence in the program at 12th months | 12 months
  Persistence assessed as the ratio between subjects followed at 12 months and subjects enrolled
Global change in traditional risk factors at 12th months | 12 months
  Assessed as the number of subjects who improved by ≥10% at least one traditional CV risk factor measure without worsening by ≥10% any other CV risk factor measure. The CV risk factors considered are: glycaemia >126 mg/dl, LDL-C >115 mg/dl, systolic blood pressure >140 mmHg and BMI >28
Global change in estimated risk at 12th months | 12 months
  Assessed as net improvement in Framingham Risk Score (number of subjects who reduced the score minus number of subjects who increased the score)

CONTACTS AND LOCATIONS:
Overall Officials: José Pablo P Werba, MD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Werba JP, Giroli MG, Simonelli N, Vigo L, Gorini A, Bonomi A, Veglia F, Tremoli E. Uptake and effectiveness of a primary cardiovascular prevention program in an underserved multiethnic urban community. Nutr Metab Cardiovasc Dis. 2022 May;32(5):1110-1120. doi: 10.1016/j.numecd.2022.01.013. Epub 2022 Jan 16. PMID 35260313